CLINICAL TRIAL: NCT03038334
Title: Magnesium Sulfate for the Improvement of Cognition in Patients With Alzheimer Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Metabolic Therapy Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR02TCR011-17
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnesium sulfate (Experimental): All participants will apply magnesium sulfate transdermally a total of 250mg equivalent to 2 mEq every four hours per day for 90 days.
  Interventions: Dietary Supplement: Magnesium sulfate

INTERVENTIONS:
Dietary Supplement: Magnesium sulfate — Transdermal application of Magnesium sulfate 250mg every four hours per day for 90 days.

SUMMARY:
This study is to examine the possible effect of supplementing Magnesium sulfate on patients with Alzheimer Disease (AD) in controlling or reducing the amount of amyloid present in the brain, and increasing cognitive ability in individuals that have amyloid deposits.

DETAILED DESCRIPTION:
Recent findings suggest magnesium may be effective in ameliorating symptoms in an Alzheimer's disease-like pathological progression by reducing Aβ-plaque, thus preventing synapse loss and memory decline in transgenic mice. Common forms include magnesium sulfate.

As a nutritional adjunct in hyperalimentation, the precise mechanism of action for magnesium is uncertain. Predominant deficiency effects are neurological, e.g., muscle irritability, clonic twitching and tremors. Hypocalcemia and hypokalemia often follow low serum levels of magnesium. While there are large stores of magnesium present intracellularly and in the bones of adults, these stores often are not mobilized sufficiently to maintain plasma levels. Parenteral magnesium therapy repairs the plasma deficit and causes deficiency symptoms and signs to cease.

To provide a comprehensive clinical evaluation of the effects of Magnesium sulfate in AD patients, this study is designed to assess the impact of magnesium sulfate on amyloid plaque to generate valuable data on clinical utility for the use of diagnostic algorithms and foundation for the development of possible treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Alzheimer's disease.
* Exhibiting an onset and progression of cognitive dysfunction during at least 3 months prior to the screening period.
* Subject or representative is willing to sign the consent for prior to enrollment into the study and to participate in all aspects of the study. Prospective subject must give verbal assent if unable to sign written consent.

Exclusion Criteria:

* Patients with neurodegenerative diseases other than Alzheimer's disease.
* Patients with cognitive dysfunction due to cerebral damage resulting from a lack of oxygen, a brain injury, etc.
* Patients with clinically significant cardiovascular disease.
* Patients with history of clinically-evident stroke.
* Patients with history of cancer in the last 5 years.
* Patients with clinically-significant systemic illness that may affect safety or completion of the study.
* Currently taking any medications that are known to interact with magnesium.
* Currently taking antibiotics as the study product may reduce the absorption of antibiotics. A washout period of 2 weeks is allowed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in amyloid deposit | Baseline to 12 weeks
  Amyloid deposit measure will mean change from baseline to 12 weeks in Florbetapir cortical-to-cerebellar ratio averaged across 6 regions of interest (frontal, temporal, parietal, anterior cingulate, posterior cingulate, and precuneus).Brain imaging focusing on the following anatomical regions: medial temporal region (including hippocampus andentorhinal cortex), prefrontal cortex, parietotemporal cortex, posterior cingulate cortex.

SECONDARY OUTCOMES:
Cognitive Function | Baseline to 12 weeks
  Composite scores for the four following cognitive areas include: 1) memory composite score 2) attention composite score 3) learning composite score 4) executive function composite score

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Haley, PhD, Principal Investigator — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: Undecided